CLINICAL TRIAL: NCT05562635
Title: Assesment of ODF ( Oral Dissolvable Film) With Long-term CBD Release in the Treatment of Temporomandibular Disorders
Brief Title: CBD (Cannabidiol) Intraoral Application and TMD (Temporomandibular Disorders)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBD (Cannabidiol)
Record Dates: First submitted 2022-08-31; First posted 2022-10-03 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-01

CONDITIONS: Temporomandibular Disorder; Myofascial Pain; Orofacial Pain; CBD; Bruxism
Keywords: temporomandibular disorder; orofacial pain; CBD; bruxism; masticatory muscles
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain; Bruxism

STUDY DESIGN:
Intervention Model Description: two groups parallel study: experimental and control group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5 % polymers with CBD application (Experimental): Bilateral application of 5% polymer gel with CBD intraorally, on the masseter muscle
  Interventions: Combination Product: 5% polymer gel with CBD application
- 10 % polymers with CBD application (Experimental): Bilateral application of 10% polymer gel with CBD intraorally, on the masseter muscle
  Interventions: Combination Product: 10% polymer gel with CBD application
- Placebo group (Placebo Comparator): Application of polymers without CBD on the masseter muscles, bilaterally
  Interventions: Combination Product: Placebo intervention

INTERVENTIONS:
Combination Product: 5% polymer gel with CBD application — Bilateral application of 5% polymer gel with CBD intraorally, on the masseter muscle
  Arms: 5 % polymers with CBD application
Combination Product: 10% polymer gel with CBD application — Bilateral application of 10% polymer gel with CBD intraorally, on the masseter muscle
  Arms: 10 % polymers with CBD application
Combination Product: Placebo intervention — Application of placebo without CBD
  Arms: Placebo group

SUMMARY:
The aim of the project is to assess the effectiveness of reducing the masseter muscles tension and hyperactivity in patients with a painful form of TMD by using polymers containing CBD compared to placebo polymers.

DETAILED DESCRIPTION:
Since the healing properties of CBD have been known for a long time, the assumption of the proposed research is to reduce the tension of the masseter muscles, reduce the bruxism index and occlusal strength, as well as reduce pain, from which patients with TMD suffer.

CBD intraoral application therapy seems promising in that field. Patients attending The Department of TMD in Zabrze, Polska will be randomly divided into two groups: experimental and placebo. sEMG activity values will be compared during 14 and 30 days therapy with polymers. the efficacy of the cannabis cream used in the study. Positive results will confirm the efficacy of CBD relaxing properties used in the study, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient agreement to participate into the research study
* Age ≥18 and ≤ 60
* Good general health,
* Temporomandibular disorder-positive RDC/TMD examination for group Ia and Ib
* Presence of all teeth (with the exception of the third molars)

Exclusion Criteria:

* Cannabis cream/ placebo cream allergy
* Hypersensitivity to substances to be used in the study
* Wounds intra oral cavity
* Addiction to cannabis
* Patients being treated with analgesic drugs and/or drugs that affect muscle function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-18 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in masseter muscle electromyographic activity- sEMG examination | 30 days
  Change in masseter muscle electromyographic activity-sEMG examination
Orofacial pain changes | 30 days
  Changes of felt pain recorded by means of VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of TMD, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walczynska-Dragon K, Grzyb A, Dawiec K, Pawlowska M, Fiegler-Rudol J, Hadzik P, Nitecka-Buchta A, Baron S. Halloysite-Assisted Delivery of Cannabidiol for the Management of Temporomandibular Pain: A Pilot Study. J Clin Med. 2025 Dec 24;15(1):145. doi: 10.3390/jcm15010145. PMID 41517391